CLINICAL TRIAL: NCT01695148
Title: Efficacy of β-carotene Biofortified Maize in Improving Vitamin A Status and Reducing the Prevalence of Vitamin A Deficiency Among Children in Rural Zambia
Brief Title: Efficacy of β-carotene Biofortified Maize in Reducing Vitamin A Deficiency Among Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Food and Nutrition Commission, Zambia (Unknown); Tropical Diseases Research Centre, Zambia (Other Government); HarvestPlus (Other); Canadian International Development Agency (Other Government); Zambia Agriculture Research Institute (Other)
Responsible Party: Principal Investigator, Keith P. West, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHU IRB 4150
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Vitamin A Deficiency; Low Serum Retinol
Keywords: beta-carotene biofortified maize; micronutrients; vitamin A; serum retinol; dark adaptation
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- White Maize Flour (Active Comparator): Children will receive 2 meals a day (~200 g of white maize flour), 6 days a week for 6 months.
  Interventions: Dietary Supplement: White Maize Flour
- β-Carotene Biofortified Maize (Experimental): Children will receive 2 meals a day (~200 g of beta-carotene biofortified maize flour), 6 days a week for 6 months.
  Interventions: Dietary Supplement: β-Carotene Biofortified Maize Flour
- Non-Intervened (No Intervention): Children will receive no food for the duration of the study, but families in this group will receive an equivalent ration of food items at the end of the trial.

INTERVENTIONS:
Dietary Supplement: β-Carotene Biofortified Maize Flour
  Arms: β-Carotene Biofortified Maize
Dietary Supplement: White Maize Flour
  Arms: White Maize Flour

SUMMARY:
The purpose of this cluster-randomized trial is to examine whether daily consumption of β-carotene biofortified maize flour can reduce the prevalence of vitamin A deficiency and improve the vitamin A status and among 4-8 year old children in rural Zambia.

DETAILED DESCRIPTION:
Vitamin A deficiency is a major public health problem in Zambia, affecting approximately 40% of young children. We aim to conduct a cluster-randomised controlled trial in the Mkushi region of rural Zambia to test whether feeding children two daily meals containing β-carotene biofortified maize flour compared to regular white maize flour-based meals for six months can reduce the prevalence of vitamin A deficiency and improve the vitamin A status among 4-8 year old children. Five hundred children in each arm will receive 2 meals a day, 6 days a week for 6 months, after which changes in serum retinol concentrations will be compared. An additional arm of 250 children, enrolled from randomly sampled clusters, will not receive the maize flour intervention but concurrently followed in order to evaluate overall effects of the maize flour feeding scheme on measures of household food security.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-8 years of age

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1228 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Increased Serum Retinol Concentration | After 6 months of feeding
  The investigators hypothesize a difference of 2.5 μg/dL or more in serum retinol among children receiving biofortified versus white maize flour-based meals. Serum retinol measures will be collected at baseline and at the end of 6 months and assessed by a High Performance Liquid Chromatography assay.
Decreased Prevalence of Vitamin A deficiency | After 6 months of feeding
  The investigators hypothesize a difference of 10% or more in the prevalence of vitamin A deficiency (i.e., serum retinol < 0.7 μmol/l) among children consuming biofortified versus white maize flour-based meals, assuming a baseline prevalence of 40%.

SECONDARY OUTCOMES:
Improved Dark Adaptation | After 6 months of Feeding
  The investigators hypothesize a difference in pupillary response to a light stimulus, as detected by dark adaptometry, in children receiving biofortified versus white maize flour-based meals.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda C Palmer, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health; Rolf Klemm, DrPH, Study Director — Johns Hopkins Bloomberg School of Public Health; Kerry J Schulze, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health; Alain Labrique, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health; Parul Christian, DrPH, Study Director — Johns Hopkins Bloomberg School of Public Health; Sucheta Mehra, MS, Study Director — Johns Hopkins Bloomberg School of Public Health; Lee Shu-Fune Wu, MS, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- JHU Office, Mkushi, Zambia

REFERENCES:
- [Background] Howe JA, Tanumihardjo SA. Carotenoid-biofortified maize maintains adequate vitamin a status in Mongolian gerbils. J Nutr. 2006 Oct;136(10):2562-7. doi: 10.1093/jn/136.10.2562. PMID 16988127
- [Background] Howe JA, Tanumihardjo SA. Evaluation of analytical methods for carotenoid extraction from biofortified maize (Zea mays sp.). J Agric Food Chem. 2006 Oct 18;54(21):7992-7. doi: 10.1021/jf062256f. PMID 17032000
- [Background] Davis C, Jing H, Howe JA, Rocheford T, Tanumihardjo SA. beta-Cryptoxanthin from supplements or carotenoid-enhanced maize maintains liver vitamin A in Mongolian gerbils ( Meriones unguiculatus) better than or equal to beta-carotene supplements. Br J Nutr. 2008 Oct;100(4):786-93. doi: 10.1017/S0007114508944123. Epub 2008 Mar 3. PMID 18312712
- [Background] Davis CR, Howe JA, Rocheford TR, Tanumihardjo SA. The xanthophyll composition of biofortified maize (Zea mays Sp.) does not influence the bioefficacy of provitamin a carotenoids in Mongolian gerbils (Meriones unguiculatus). J Agric Food Chem. 2008 Aug 13;56(15):6745-50. doi: 10.1021/jf800816q. Epub 2008 Jul 11. PMID 18616269
- [Background] Muzhingi T, Gadaga TH, Siwela AH, Grusak MA, Russell RM, Tang G. Yellow maize with high beta-carotene is an effective source of vitamin A in healthy Zimbabwean men. Am J Clin Nutr. 2011 Aug;94(2):510-9. doi: 10.3945/ajcn.110.006486. Epub 2011 Jun 29. PMID 21715509
- [Derived] Healy K, Palmer AC, Barffour MA, Schulze KJ, Siamusantu W, Chileshe J, West KP Jr, Labrique AB. Nutritional Status Measures Are Correlated with Pupillary Responsiveness in Zambian Children. J Nutr. 2018 Jul 1;148(7):1160-1166. doi: 10.1093/jn/nxy069. PMID 29924320
- [Derived] Palmer AC, Craft NE, Schulze KJ, Barffour M, Chileshe J, Siamusantu W, West KP Jr. Impact of biofortified maize consumption on serum carotenoid concentrations in Zambian children. Eur J Clin Nutr. 2018 Feb;72(2):301-303. doi: 10.1038/s41430-017-0054-1. Epub 2018 Jan 10. PMID 29321687
- [Derived] Barffour MA, Schulze KJ, Coles CL, Chileshe J, Kalungwana N, Arguello M, Siamusantu W, Moss WJ, West KP Jr, Palmer AC. High Iron Stores in the Low Malaria Season Increase Malaria Risk in the High Transmission Season in a Prospective Cohort of Rural Zambian Children. J Nutr. 2017 Aug;147(8):1531-1536. doi: 10.3945/jn.117.250381. Epub 2017 Jul 12. PMID 28701387
- [Derived] Palmer AC, Healy K, Barffour MA, Siamusantu W, Chileshe J, Schulze KJ, West KP Jr, Labrique AB. Provitamin A Carotenoid-Biofortified Maize Consumption Increases Pupillary Responsiveness among Zambian Children in a Randomized Controlled Trial. J Nutr. 2016 Dec;146(12):2551-2558. doi: 10.3945/jn.116.239202. Epub 2016 Oct 19. PMID 27798345
- [Derived] Palmer AC, Siamusantu W, Chileshe J, Schulze KJ, Barffour M, Craft NE, Molobeka N, Kalungwana N, Arguello MA, Mitra M, Caswell B, Klemm RD, West KP Jr. Provitamin A-biofortified maize increases serum beta-carotene, but not retinol, in marginally nourished children: a cluster-randomized trial in rural Zambia. Am J Clin Nutr. 2016 Jul;104(1):181-90. doi: 10.3945/ajcn.116.132571. Epub 2016 May 11. PMID 27169838